CLINICAL TRIAL: NCT03519880
Title: A Pilot Study of the Utility of 3D Printed Masks for ALS Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 research restrictions
Sponsor: University of Michigan (Other)
Collaborators: ALS Association (Other)
Responsible Party: Principal Investigator, Stephen Goutman, Assistant Professor of Neurology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00112433
Record Dates: First submitted 2018-04-16; First posted 2018-05-09 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis, non-invasive ventilation, mask, custom, 3D-printing
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: All trial enrollees will receive the custom-designed 3D printed non-invasive ventilation mask interface.
Masking Description: There is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Custom Mask Interface (Experimental): Patients use a custom mask interface for one month with an option to use for a year if it performs better than a commercial mask.
  Interventions: Device: Custom Mask Interface

INTERVENTIONS:
Device: Custom Mask Interface — Subjects enrolled in the study will received a custom designed, 3D printed, non-invasive ventilation mask interface.

SUMMARY:
Non-invasive ventilation (NIV) is an important therapy for patients with a number of neurological diseases. Specifically, NIV has been shown to be an effective treatment for people with amyotrophic lateral sclerosis (ALS, also known as Lou Gehrig's disease), which is a fatal, non-curable, progressive disease of the motor neurons. However, due to changes in facial structure associated with the disease, many ALS patients find that traditional NIV masks don't fit well. In this study, investigators will perform a feasibility study on NIV mask interfaces which are custom designed for each ALS patient and then manufactured via 3D printing.

DETAILED DESCRIPTION:
Non-invasive ventilation (NIV) is an important therapy for patients with a number of neurological diseases. Specifically, for amyotrophic lateral sclerosis (ALS)--a fatal, non-curable, progressive disease of the motor neurons--NIV represents one of the most effective treatments with a survival benefit of greater than 1 year. Despite this survival advantage, and the corresponding improvement in Quality of Life (QoL), compliance with NIV can be poor. Factors contributing to poor compliance to NIV include bulbar onset disease and mask leaks. In addition to reduced adherence to therapy, elevated mask leaks can compromise the pressure adjustment algorithm in average volume assured pressure support (AVAPS) ventilation, a commonly used mode of bilevel (positive airway pressure) PAP therapy in ALS. In an effort to increase NIV compliance in subjects with neurological conditions, and specifically ALS, investigators hypothesize that a better fit achieved through 3D printed NIV mask interfaces may improve utilization by decreasing mask leaks, decreasing the required delivery pressures and improving compliance with therapy. Investigators therefore propose a feasibility study to investigate the use of 3D printing to manufacture customized NIV mask interfaces for subjects with ALS who encounter difficulty using NIV because of poorly fitting mask interfaces despite exhausting available commercial mask options.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 18
2. Ability to communicate in English
3. Diagnosis of ALS
4. Subject followed in the ALS Clinic at University of Michigan
5. Current use of NIV.
6. Problematic mask leak defined as one of the following:

   A. A clinical complaint of mask leak impeding use of PAP AND PAP use <6 hours per night AND/OR B. Average percentage of the night in large leak on download of >10% (AVAPS)
7. At least 1 month of NIV use

Exclusion Criteria:

1. Subjects successfully using a commercially available mask without objective or subjective leak with good compliance (average use >6 hours per night)
2. Silicone allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Average number of hours the custom NIV mask interface is used per night | 1 month
  Average number of hours the custom NIV mask interface is used per night
Leak parameters from device | 1 month
  Average minutes in large leak or leak measured from the device in liters per minute and averaged over the month
Tidal volume measurements | 1 month
  (average measured tidal volume/average set tidal volume)*100%

SECONDARY OUTCOMES:
Interviews with subjects regarding their experience with the custom mask Qualitative assessment of custom NIV mask efficacy | 1 month
  Interviews with subjects regarding their experience with the custom mask

OTHER OUTCOMES:
ALS Depression Inventory-12 (ADI-12) | 1 month
  Depression Scale. Scales: For each question, the following is selected: "I fully agree", "I agree", "I don't agree", "I do not agree at all"
ALS Functional Rating Scale, Revised (ALSFRS-R) | 1 month
  Functional Rating Scale. Scales: Customized for each question, but 4 is the maximum and generally means 'normal', and 0 represents significant impairment.
ALS Specific Quality of Life-20 (ALSSQOL20) | 1 month
  Quality of Life Scale. Scales: For each question, 1-10 is selected, where 10 means "extremely" and 0 means "not at all".
Epworth Sleepiness Scale (ESS) | 1 month
  Sleepiness Scale. Scales: 3 means "high chance of dozing", 2 means "moderate chance of dozing", 1 means "slight chance of dozing", and 0 means "would never doze".
PROMIS Neuro-Quality of Life Fatigue Scale | 1 month
  Fatigue Scale. Scales: For each question, "Always" (5), "Often" (4), "Sometimes" (3), "Rarely" (2), and "Never" (1) is selected.
PROMIS Neuro-Quality of Life Sleep Disturbance Scale | 1 month
  Sleep Disturbance Scale. Scales: For each question, "Always" (5), "Often" (4), "Sometimes" (3), "Rarely" (2), and "Never" (1) is selected.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A Goutman, MD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Medicine, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No